CLINICAL TRIAL: NCT00139620
Title: An Open-Label Study to Characterize the Pharmacokinetic Parameters of Erlotinib (Tarceva®, OSI-774) in Cancer Patients With Advanced Solid Tumors, With Adequate and Moderately Impaired Hepatic Function
Brief Title: A Pharmacokinetic Study of Erlotinib in Cancer Patients With Advanced Solid Tumors, With Adequate and Moderately Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Organization: Astellas Pharma Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-104; 2006-002363-59 (EudraCT Number)
Record Dates: First submitted 2005-08-25; First posted 2005-08-31 (Estimated); Last update posted 2018-02-08 (Actual); Status verified 2015-06

CONDITIONS: Advanced Solid Tumors
Keywords: advanced cancer, solid tumor
MeSH Terms: interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva, erlotinib, OSI-774

SUMMARY:
This is a multicenter, open-label, 2-arm study comparing erlotinib exposure in cancer patients with adequate hepatic function versus cancer patients with moderate hepatic impairment. All patients will receive a single 150 mg dose of erlotinib on Day 1 followed by 96 hours of plasma sampling for PK and protein binding studies. Patients may then enter the maintenance phase of the study and continue to receive erlotinib until disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced solid tumor (measurable or nonmeasurable) that is potentially responsive to erlotinib or for which no effective therapy is available,
* Cohort 1: Adequate hepatic function: bilirubin <= ULN, ALT (SGPT) and AST (SGOT) <= 1.5 x ULN or Cohort 2: Moderate hepatic function: 7-9 as assessed by the Child-Pugh System, ECOG Performance Status 0-2
* Life expectancy >= 12 weeks,
* Prior radiation permitted provided that 4 weeks (or 2 weeks for palliative radiation) has elapsed and patients have recovered from acute toxic effects of radiotherapy,
* Prior chemotherapy permitted provided that 4 weeks has elapsed and patients have recovered from acute toxic effects of chemotherapy,
* Adequate hematopoietic and renal function: ANC >= 1.5 x 10^9/L, platelets >= 75 x 10^9/L, and creatinine <= 1.5 x ULN,

Exclusion Criteria:

* Use of tobacco or nicotine-containing products within 4 weeks of Day 1 and while on study,
* Use of a CYP3A4 inhibitor or inducer within 14 days prior to Day 1 and until Day 5,
* Use of a warfarin-derivative anticoagulant within 14 days prior to Day 1 and until Day 5,
* Encephalopathy >= grade 2,
* Significant history of cardiac disease unless well-controlled,
* Active or uncontrolled infections or serious illnesses or medical conditions that could interfere with the patient's ongoing participation,
* Concurrent anticancer therapy or any other investigational agents within 4 weeks of Day 1 and while on study,
* Symptomatic brain metastases that are not stable, require steroids, are potentially life-threatening, or that have required radiation within the last 4 weeks,
* Gastro-intestinal abnormalities, including inability to take oral medication, requirement for IV alimentation, active peptic ulcer or prior surgical procedures affecting absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-08-22 (Actual); Primary Completion 2007-06-25 (Actual); Study Completion 2007-06-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Premiere Oncology, Santa Monica, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Mayo Clinic, Rochester, Minnesota
  - UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
- The Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=55